CLINICAL TRIAL: NCT00288925
Title: Phase Ib/IIa, to Evaluate the Safety and Pharmacokinetics of Z-360 in Subjects With Unresectable Advanced Pancreatic Cancer in Combination With Gemcitabine Treatment
Brief Title: Z-360 in Unresectable Advanced Pancreatic Cancer in Combination With Gemcitabine Treatment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zeria Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01010106E
Record Dates: First submitted 2006-02-06; First posted 2006-02-08 (Estimated); Last update posted 2009-06-01 (Estimated); Status verified 2009-05

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Z-360

INTERVENTIONS:
Drug: Z-360

SUMMARY:
To evaluate the safety of two doses of Z-360 with Gemcitabine administration for subjects with unresectable advanced pancreatic cancer in order to determine the optimal dosage for PhaseII study

ELIGIBILITY:
Inclusion Criteria:

* Subjects with unresectable locally advanced or metastatic pancreatic cancer
* KPS > 70%
* Life expectancy of at least 3 months

Exclusion Criteria:

* received previous chemotherapy for the current indication
* received previous radiotherapy for the current indication
* Currently receiving chemotherapy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-09; Primary Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Safety, Pharmacokinetics

SECONDARY OUTCOMES:
Tumour shrinkage, Tumour objective response rate

CONTACTS AND LOCATIONS:
Overall Officials: Tim Meyer, PhD, MD, Principal Investigator — Royal Free Hospital NHS Foundation Trust
Locations (1):
- Royal Free Hospital, London, United Kingdom